CLINICAL TRIAL: NCT04057534
Title: Investigating Neurobiological Mechanisms of Chess as an Add-On Treatment Against Substance Use Disorder
Brief Title: Neurobiological Mechanisms of Chess as an Add-On Treatment Against SUD
Acronym: Chess_SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chess_SUD
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Substance Use Disorders
Keywords: Alcohol Dependence; Alcoholism; Craving; Cognitive Change; cognitive remediation; Chess based cognitive training; Working Memory; Decision Making; Executive Control; Chess; fMRI; Nicotine use disorder; Tobacco use disorder
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Tobacco Use Disorder | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CB-CRT AUD group (Experimental): experimental group AUD: patients receive standard clinical therapy and an add-on chess based - cognitive remediation treatment (CB-CRT)
  Interventions: Behavioral: Standard therapy for AUD plus Chess-based cognitive treatment
- Control group AUD (Active Comparator): control group: patients with AUD receive standard clinical therapy
  Interventions: Behavioral: Standard therapy for AUD
- CB-CRT TUD group (Experimental): experimental group TUD: patients receive standard smoking cessation therapy and an add-on CB-CRT
  Interventions: Behavioral: Standard smoking cessation therapy for TUD plus Chess-based cognitive treatment
- Control group TUD (Active Comparator): control group: patients with TUD receive standard smoking cessation therapy
  Interventions: Behavioral: Standard therapy for TUD

INTERVENTIONS:
Behavioral: Standard therapy for AUD plus Chess-based cognitive treatment — Behavioral: standard AUD Cognitive Behavioral Therapy (CBT) in Clinical setting.
  Patients who voluntarily submit to enter a qualified detoxification treatment program will be examined, either in-patient, out-patient, or in a day-clinic setting at the Department of Addictive Behaviour and Addiction Medicine. Additional, the experimental group receives chess based cognitive remediation treatment (CB-CRT) for 1,5 hours three times a week. The tasks of the treatment were created by our cooperation partner, the psychologist Juan Antonio Montero. He is currently successfully applying this battery as an add-on therapy. The training battery is designed to strengthen cognitive functioning in specific domains such as short-term memory, focal attention, selective attention, pattern recognition, visuospatial abilities, metacognition and also inhibition.
  Arms: CB-CRT AUD group
Behavioral: Standard therapy for AUD — Behavioral: standard AUD Cognitive Behavioral Therapy (CBT) in Clinical setting. Patients who voluntarily submit to enter a qualified detoxification treatment program will be examined, either in-patient, out-patient, or in a day-clinic setting at the Department of Addictive Behaviour and Addiction Medicine.
  Arms: Control group AUD
Behavioral: Standard smoking cessation therapy for TUD plus Chess-based cognitive treatment — Behavioral: standard smoking cessation therapy for TUD in group therapy setting.
  Patients who voluntarily submit to enter a qualified smoking cessation program will be examined in an out-patient setting at the Department of Addictive Behaviour and Addiction Medicine. They receive a six-week standard therapy (one 1,5 hours group therapy per week). Additional, the experimental group receives chess based cognitive remediation treatment (CB-CRT) for 1,5 hours three times a week. The tasks of the treatment were created by our cooperation partner, the psychologist Juan Antonio Montero. He is currently successfully applying this battery as an add-on therapy. The training battery is designed to strengthen cognitive functioning in specific domains such as short-term memory, focal attention, selective attention, pattern recognition, visuospatial abilities, metacognition and also inhibition.
  Arms: CB-CRT TUD group
Behavioral: Standard therapy for TUD — Behavioral: standard smoking cessation therapy for TUD in group therapy setting.
  Patients who voluntarily submit to enter a qualified smokind cessation program will be examined in an out-patient setting at the Department of Addictive Behaviour and Addiction Medicine. They receive a six-week standard therapy (one 1,5 hours group therapy per week). Additional, the experimental group receives chess based cognitive remediation treatment (CB-CRT) for 1,5 hours three times a week.
  Arms: Control group TUD

SUMMARY:
Neurobiological and neuropsychological approaches to investigate the potential mechanism of action of chess as an add-on therapy (chess based - cognitive remediation treatment, CB-CRT) to reduce cognitive deficits in individuals with alcohol use disorder (AUD) or tobacco use disorder (TUD).

DETAILED DESCRIPTION:
The study aims to investigate the potential mechanism of action of chess as a "chess based - cognitive remediation treatment, CB-CRT" to reduce cognitive deficits in individuals with substance use disorder (SUD) seeking treatment using neurobiological and neuropsychological approaches. Furthermore, it will be assessed whether this chess intervention has a generalized positive effect on short-term abstinence. Interestingly, the functional domains and associated underlying neuronal networks observed to be affected in individuals with SUD overlap significantly with those that could be strengthened by chess-based cognitive training or formal chess. Specifically, strengthening of cortical control regions (dorsolateral prefrontal cortex, DLPFC) and brain areas relevant for decision-making (orbitofrontal cortex, OFC) could prevent future relapse. Therefore, chess as an add-on therapy to complement other standard treatments of SUD could lead to improved therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* severe alcohol (AUD) or tabacco use disorder (SUD) according to DSM-5
* abstinence from alcohol for at least 72 hours (AUD)
* sufficient ability to communicate with investigators and answer questions in both written and verbal format
* ability to provide fully informed consent and to use self-rating scales
* main diagnosis AUD: inpatient or outpatient treatment in our clinic
* main diagnosis TUD: participation in 6 weeks smoking cessation treatment
* Normal or corrected to normal vision
* Signed consents for data security

Exclusion Criteria:

* severe internal, neurological, and/or psychiatric comorbidities; other Axis I mental disorders other than TUD according to ICD-10 and DSM 5 (except for other substance use disorders - if AUD or TUD is still the main diagnosis -, ADHD, remitted depression, mild or moderate depression, adjustment disorder, generalized anxiety disorder, phobias, panic disorder or other mild or moderate personality disorders) in the last 12 months
* Severe withdrawal symptoms (CIWA-Ar > 7; Sullivan et al. 1989)
* alcohol intoxication (>0‰)
* history of brain injury
* severe cognitive impairments
* common exclusion criteria for MRI (e.g. metal, claustrophobia, pregnancy)
* suicidality or endangerment of others
* positive Covid-19 screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
change in neural alcohol cue-reactivity | 2 time points: before and after 6 weeks chess-based cognitive training
  fMRI alcohol cue-reactivity task (Vollstädt-Klein et al. 2010)
change in neural tobacco cue-reactivity | 2 time points: before and after 6 weeks chess-based cognitive training
  fMRI tobacco cue-reactivity task (Vollstädt-Klein et al. 2011)
change in neural correlates of inhibition | 2 time points: before and after 6 weeks chess-based cognitive training
  fMRI stop-signal task (Whelan et al. 2012)
substance use (alcohol consumption and tabacco use) | 3 months follow-up after the end of treatment
  self-report
change in neural working memory processes | 2 time points: before and after 6 weeks chess-based cognitive training
  fMRI working memory task "N-back" (Charlet et al. 2014)
Change in working memory capacity | 2 time points: before and after 6 weeks SCP
  working memory capacity measured by letter-number sequencing task of the [Wechsler Memory Scale (Kent 2013)]; raw values will be transformed to IQ-like scales (mean 100, SD 15); the higher the value, the higher the working memory capacity
Change in impulsivity | 3 time points: before and after 6 weeks SCP plus after 3 months
  impulsivity measured with BIS scale [Barratt impulsiveness scale (Patton et al. 1995)];range 15-60; total score will be used; high values represent high impulsivity
Change in decision-making | 2 time points: before and after 6 weeks SCP
  [Iowa Gambling Task (Bechara et al. 1994)]
Change in mental flexibility | 2 time points: before and after 6 weeks SCP
  [Dimensional Change Card Sort (Zelazo et al. 2014)]
Change in attentional capacity | 2 time points: before and after 6 weeks SCP
  [d2 Test of Attention (Brickenkamp 2002)].

SECONDARY OUTCOMES:
change in functional connectivity within the salience network (SN) and executive control network (ECN) | 2 time points: before and after 6 weeks therapy and chess-based cognitive training
  [measured with fMRI]

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Yes
For protection of personal rights, and due to the sensitivity of the clinical and neuroimaging data, data will not be made publicly available. Upon direct request by other researchers and in mutual agreements (e.g., regarding data protection), anonymized data can be made available. Upon request, analysis procedures and codes will be shared with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: After publication
Access Criteria: Upon request by researchers or institution following the current data protection laws.

REFERENCES:
- [Background] Adinoff B. Neurobiologic processes in drug reward and addiction. Harv Rev Psychiatry. 2004 Nov-Dec;12(6):305-20. doi: 10.1080/10673220490910844. PMID 15764467
- [Background] Fauth-Buhler M, de Rover M, Rubia K, Garavan H, Abbott S, Clark L, Vollstadt-Klein S, Mann K, Schumann G, Robbins TW. Brain networks subserving fixed versus performance-adjusted delay stop trials in a stop signal task. Behav Brain Res. 2012 Nov 1;235(1):89-97. doi: 10.1016/j.bbr.2012.07.023. Epub 2012 Jul 20. PMID 22820235
- [Result] Amidzic O, Riehle HJ, Fehr T, Wienbruch C, Elbert T. Pattern of focal gamma-bursts in chess players. Nature. 2001 Aug 9;412(6847):603. doi: 10.1038/35088119. No abstract available. PMID 11493907
- [Result] Atherton M, Zhuang J, Bart WM, Hu X, He S. A functional MRI study of high-level cognition. I. The game of chess. Brain Res Cogn Brain Res. 2003 Mar;16(1):26-31. doi: 10.1016/s0926-6410(02)00207-0. PMID 12589885
- [Result] Bates ME, Buckman JF, Nguyen TT. A role for cognitive rehabilitation in increasing the effectiveness of treatment for alcohol use disorders. Neuropsychol Rev. 2013 Mar;23(1):27-47. doi: 10.1007/s11065-013-9228-3. Epub 2013 Feb 15. PMID 23412885
- [Result] Blasco-Fontecilla H, Gonzalez-Perez M, Garcia-Lopez R, Poza-Cano B, Perez-Moreno MR, de Leon-Martinez V, Otero-Perez J. Efficacy of chess training for the treatment of ADHD: A prospective, open label study. Rev Psiquiatr Salud Ment. 2016 Jan-Mar;9(1):13-21. doi: 10.1016/j.rpsm.2015.02.003. Epub 2015 Apr 22. English, Spanish. PMID 25911280
- [Result] Demily C, Cavezian C, Desmurget M, Berquand-Merle M, Chambon V, Franck N. The game of chess enhances cognitive abilities in schizophrenia. Schizophr Res. 2009 Jan;107(1):112-3. doi: 10.1016/j.schres.2008.09.024. Epub 2008 Nov 7. No abstract available. PMID 18995990
- [Result] Fattahi F, Geshani A, Jafari Z, Jalaie S, Salman Mahini M. Auditory memory function in expert chess players. Med J Islam Repub Iran. 2015 Oct 6;29:275. eCollection 2015. PMID 26793666
- [Result] Goncalves PD, Ometto M, Bechara A, Malbergier A, Amaral R, Nicastri S, Martins PA, Beraldo L, dos Santos B, Fuentes D, Andrade AG, Busatto GF, Cunha PJ. Motivational interviewing combined with chess accelerates improvement in executive functions in cocaine dependent patients: a one-month prospective study. Drug Alcohol Depend. 2014 Aug 1;141:79-84. doi: 10.1016/j.drugalcdep.2014.05.006. Epub 2014 May 24. PMID 24913200
- [Result] Onofrj M, Curatola L, Valentini G, Antonelli M, Thomas A, Fulgente T. Non-dominant dorsal-prefrontal activation during chess problem solution evidenced by single photon emission computerized tomography (SPECT). Neurosci Lett. 1995 Oct 6;198(3):169-72. doi: 10.1016/0304-3940(95)11985-6. PMID 8552313
- [Result] Vollstadt-Klein S, Wichert S, Rabinstein J, Buhler M, Klein O, Ende G, Hermann D, Mann K. Initial, habitual and compulsive alcohol use is characterized by a shift of cue processing from ventral to dorsal striatum. Addiction. 2010 Oct;105(10):1741-9. doi: 10.1111/j.1360-0443.2010.03022.x. PMID 20670348
- [Result] Lally N, Huys QJM, Eshel N, Faulkner P, Dayan P, Roiser JP. The Neural Basis of Aversive Pavlovian Guidance during Planning. J Neurosci. 2017 Oct 18;37(42):10215-10229. doi: 10.1523/JNEUROSCI.0085-17.2017. Epub 2017 Sep 18. PMID 28924006
- [Derived] Gerhardt S, Lex G, Holzammer J, Karl D, Wieland A, Schmitt R, Recuero AJ, Montero JA, Weber T, Vollstadt-Klein S. Effects of chess-based cognitive remediation training as therapy add-on in alcohol and tobacco use disorders: protocol of a randomised, controlled clinical fMRI trial. BMJ Open. 2022 Sep 6;12(9):e057707. doi: 10.1136/bmjopen-2021-057707. PMID 36691127